CLINICAL TRIAL: NCT06578143
Title: Effects of Synbiotics on Obesity and Obesity-related Parameters
Brief Title: Effects of Synbiotics on Obesity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leeuwenhoek Laboratories Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LL-IRB-2402
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Other: Placebo
- Synbiotics (Experimental)
  Interventions: Other: Synbiotics

INTERVENTIONS:
Other: Placebo — Placebo is administered in capsules (500 mg each). Participants are instructed to take the capsules twice daily, with two capsules per dose, after meals. The duration of the intervention is 6 weeks.
  Arms: Control
Other: Synbiotics — Synbiotics is administered in capsules (500 mg each). Participants are instructed to take the capsules twice daily, with two capsules per dose, after meals. The duration of the intervention is 6 weeks.
  Arms: Synbiotics

SUMMARY:
Synbiotics are a combination of probiotics and prebiotics that can promote the survival of probiotics in the gut. Probiotics utilize prebiotics to produce various metabolites beneficial to human health, such as short-chain fatty acids. The purpose of this trial is to evaluate the impact of a synbiotics product developed by Leewenhoek Laboratories Co., Ltd., on human obesity and its related biomarkers. Participants will be randomly assigned to either the experimental group or the control group in a double-blind trial. The intervention involves the experimental group taking the synbiotics product twice daily, two capsules per dose, after meals for six weeks. The control group will take an equal amount of placebo daily. During the trial, participants' body weight will be recorded weekly, and their body weight, waist circumference, hip circumference, body fat composition, and skeletal muscle mass will be measured before and after the intervention. Additionally, fasting blood samples and blood samples collected at 30, 60, 90, and 120 minutes after consuming the nutritional supplements will be analyzed. The study will compare body fat percentage, body weight, BMI, waist circumference, hip circumference, skeletal muscle mass, and obesity-related biomarkers in blood between the experimental and control groups. The trial results will be used to assess the efficacy of the synbiotics product in improving obesity and its related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60 years.
* Body weight ≥ 50 kg.
* Body Mass Index (BMI) ≥ 24.
* Body fat percentage ≥ 30% for females or ≥ 25% for males.
* Waist circumference ≥ 80 cm for females or ≥ 90 cm for males.
* No remarkable medical history within the past six months.
* Willing to comply with the nutritional instructions during the study period.
* Willing to report body weight once a week.
* Willing to report dietary and activity records.
* Willing to comply with the instruction of "not using" other products containing probiotics or enzymes (excluding yogurt and yogurt drinks).
* Willing to sign Clinical Trial Informed Consent Form before the trial.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Without statutory notifiable diseases, including HIV, syphilis, hepatitis B, hepatitis C, etc.
* Judged by a physician to have "secondary obesity" (obesity caused by endocrine disorders or metabolic abnormalities).
* Presence of endocrine disorders, hypertension, diabetes, cerebrovascular diseases, cardiovascular diseases, liver diseases, kidney diseases, gastrointestinal diseases, or mental disorders.
* Currently taking medications for lipid-lowering, blood sugar control, or weight loss.
* Currently taking antibiotic-related medications.
* Determined unsuitable for participation in this trial by a physician.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Body fat percentage | Up to six weeks
  The difference in body fat percentage between experimental group and control group.